CLINICAL TRIAL: NCT02849678
Title: A Comparison of Lidocaine Versus Ropivacaine for Bilateral Continuous Thoracic Paravertebral Nerve Blocks for Post-bowel Surgery Analgesia
Brief Title: A Pain Study Comparing Two Commonly Used Medications to Treat Pain After Bowel Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Vice Chair of Clinical Research, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO07080230
Record Dates: First submitted 2016-03-22; First posted 2016-07-29 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain; Bowel Surgery; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine will be infused through a catheter placed in the thoracic paravertebral space to block the transmission of pain signals at the level of the spinal nerves from the abdominal incision.
  At a concentration of 0.5%, Lidocaine has been deemed safe to use for peripheral nerve blocks and analgesia.Compared to ropivacaine, lidocaine is shorter-acting, less cardiotoxic, and safer to use.
  Interventions: Drug: Lidocaine
- Ropivacaine (Active Comparator): Ropivacaine is a local anesthetic used as the standard drug in paravertebral nerve blocks at our institution. It is also used in other nerve block infusions at our hospital and institutions across the country. It will be used as the standard drug to which lidocaine is compared.
  Ropivacaine has been safely used in the paravertebral nerve blocks at our institution for several years.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 0.5% Ropivacaine will be infused through a catheter placed in the thoracic paravertebral space to block the transmission of pain signals at the level of the spinal nerves from the abdominal incision. It is the local anesthetic used as the standard drug in paravertebral nerve blocks at our institution. It is also used in other nerve block infusions at our hospital and institutions across the country. It will be used as the standard drug to which lidocaine is compared.
  Other Names: Naropin®; Ropivacaine hydrochloride
  Arms: Ropivacaine
Drug: Lidocaine — Lidocaine will be infused through a catheter placed in the thoracic paravertebral space to block the transmission of pain signals at the level of the spinal nerves from the abdominal incision.
  At a concentration of 0.5%, Lidocaine has been deemed safe to use for peripheral nerve blocks and analgesia. There are several studies to support this as listed in the references. Compared to ropivacaine, lidocaine is shorter-acting, less cardiotoxic, and safer to use.
  Other Names: Xylocaine
  Arms: Lidocaine

SUMMARY:
This research study is testing whether the local anesthetic lidocaine is as effective as ropivacaine for post-operative pain control in continuous thoracic paravertebral nerve blocks. Ropivacaine and Lidocaine are FDA-approved drugs that has been successfully used in this hospital for post-operative pain control for the past few years, thus has become the standard drugs used for this nerve block. Lidocaine has numerous potential advantages over ropivacaine, such as faster onset of action, better safety profile and greater anti-inflammatory action. Catheters placed near both sides of a patient's spine for postoperative pain control are called thoracic paravertebral nerve blocks and are a part of routine care. Through those catheters, a "numbing" medication, or local anesthetic, to block the transmission of pain from the surgical incision to the spinal cord, thus reducing pain. The research part of the study is whether subjects will receive either the local anesthetic lidocaine or ropivacaine. The goal of this study is to determine whether the lidocaine controls pain better and facilitates a faster recovery after abdominal surgery than ropivacaine.

In this research study, the investigators will compare patient-reported pain scores, any additional pain medication requirements for adequate pain control, time it takes for bowel function to return to normal following surgery, as well as the incidence of any side effects, such as numbness and weakness, subjects may experience between those receiving lidocaine versus those receiving ropivacaine. The investigators will screen 100 patients and enroll 60 subjects into this study.

DETAILED DESCRIPTION:
After determining eligibility, subjects will be enrolled in one of the two study groups on the day of surgery using a sealed envelope determined by a computer-generated list that made assignments randomly based on enrollment number. The study groups are defined as:

Study group: Lidocaine 0.25%(L) 32 patients Control group: Ropivacaine 0.2%(R) 32 patients

Paravertebral nerve block catheter placement and activation:

After standard monitors and supplemental oxygen are applied, the patient will be placed in a sitting position. The two points of needle entry will be marked on the skin corresponding to each of the bilateral paravertebral catheter placements. The thoracic spine level will be at the anatomic level corresponding to the midpoint of the incision as determined by the surgeon preoperatively (range T7 to T11). The needle entry sites will be 2.5 cm lateral on each side of the midpoint of the spinous process of the corresponding thoracic vertebrae. The area will be prepared and draped in a sterile fashion, and 1% lidocaine infiltrated subcutaneously at each point of anticipated needle entry. For each of the two catheter placements, a sterile 18 gauge Tuohy needle (B. Braun Medical, Inc., Perifix Continuous Epidural Anesthesia Set, Product Code CE18T) will be introduced perpendicularly to the skin until the transverse process is encountered, and the depth to the skin will be noted. The needle will then be readjusted in a caudad direction and inserted inferior to the corresponding transverse process to a depth approximately 1 cm deep to the transverse process. After final needle placement, a hanging drop technique will be used to rule out intrapleural placement while the patient inhales and exhales deeply. Next 5 mL of 0.5% Ropivacaine will be injected incrementally through each needle after negative aspiration, followed by insertion of the nerve block catheter to a depth 5 cm beyond the tip of the needle. An additional 10 mL of 0.5% Ropivacaine will then be injected in 5 mL increments with negative aspiration in between, through each catheter yielding a total activation dose of 15 ml of 0.5% Ropivacaine on each side. The catheters will be secured with Steri-strips and a transparent occlusive dressing. Vital signs will be monitored by the nurse at regular intervals until the patient is taken to the operating room.

Postoperative Management:

Post Anesthesia Care Unit (PACU):

Following routine intraoperative general anesthesia care, management in the post-anesthesia care unit will follow the standard of care for colorectal surgery. Bilateral paravertebral infusions of ropivacaine 0.2% or lidocaine 0.25% will be started at 7 mL/hr on each side for the patients depending which to group they were randomized. The patients in both groups will also be given access to PCA dilaudid (0.2 mg bolus, 8 min lockout, no basal infusion, no 1-hour limit) once verbal pain score is ≤4. Additional pain relief is available via nurse-administered 10 mL/hour boluses of ropivacaine 0.2% or lidocaine 0.25% via the catheter pumps (5 mL each side for paravertebral group).This will be continued until the patient is able to tolerate oral pain medication. A single IV bolus of ketorolac at 7.5 mg will be available for additional pain management. Patient reported pain scores and total analgesic requirements will be recorded. Once adequate analgesia is established without any signs of adverse effects from the nerve blocks, the patients will be transferred to a hospital floor bed.

Floors:

After discharge from the PACU, additional pain relief is available via nurse-administered 3 mL boluses of local anesthetic via the catheter pumps (3 mL each side for paravertebral group) given no more than hourly. In addition, nurse-administered intravenous boluses of dilaudid 0.3 mg every 30 minutes as needed up to 2 doses while the patient has PCA, and 0.8-1 mg every hour as needed up to 4 doses in 2 hours once the patient is taking oral pain therapy and is off the PCA. All patients will be assessed daily by members of the acute interventional perioperative pain service. Also, a member of the acute pain service will be on-call 24 hours if inadequate pain control or side effects arise. The infusion rates via the paravertebral catheters may be adjusted at the discretion of the pain service up to a rate of 10 mL/hr of either lidocaine 0.25% or ropivacaine 0.2% on each side (standard infusion rate used at UPMC). The PCA dose may be adjusted as deemed necessary by the acute pain team in order provide adequate analgesia. In addition 7.5mg IV of ketorolac may be administered every 6 hours for the first 48 hours. Once the patient is able to tolerate oral liquids as determined by the surgeon, the PCA will be discontinued and oxycodone 5 mg available to the patient every 4 hours as needed for mild-moderate pain or oxycodone 10 mg every 6 hours as needed for severe pain. These doses may be adjusted as necessary by the pain service. All paravertebral catheters will be stopped and removed on the day after the patient has his/her first bowel movement or post-operative day #4, whichever occurs first. Pain scores collected by the nurses and supplemental analgesic requirements will be the data points for this study. Also, return of flatus and first bowel movement as documented in the AIPPS and surgery team's daily round notes will be recorded during the length of the hospitalization respectively.

For each patient, the investigators collected numerical rating scores (NRS) for pain at rest and during movement at baseline, at postanesthesia care unit discharge, at 24 hours and 48 hours after the end of surgery,

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III subjects
* Ages 18-80 years
* Weight between 60 and 110 Kg
* At least 60in (152cm) tall
* Scheduled for elective open colonic surgery at UPMC Presbyterian Shadyside Hospital in Pittsburgh, Pennsylvania

Exclusion Criteria:

* Age younger than 18 years or older than 80 years
* Any contraindication to the placement of bilateral thoracic paravertebral catheters
* American Society of Anesthesiologists physical status IV or greater
* Chronic painful conditions
* Preoperative opioid use
* Coagulation abnormalities or patients who are expected to be on therapeutic anticoagulants postoperatively
* Allergy to any of the drugs/agents used study protocol
* Personal or family history of malignant hyperthermia
* Serum creatinine greater than 1.3 g/dl
* Pregnancy
* Having an altered mental status (not oriented to place, person, or time)
* Emergency surgery and those with sepsis, unstable angina, congestive heart disease, valvular heart disease, and severe COPD
* Patient's inability to provide adequate informed consent
* Non-english speaking
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-01; Primary Completion 2013-11 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Fanelli, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
This data has been published.

REFERENCES:
- [Result] Ghisi D, Fanelli A, Jouguelet-Lacoste J, La Colla L, Auroux AS, Chelly JE. Lidocaine versus ropivacaine for postoperative continuous paravertebral nerve blocks in patients undergoing laparoscopic bowel surgery: a randomized, controlled, double-blinded, pilot study. Local Reg Anesth. 2015 Sep 14;8:71-7. doi: 10.2147/LRA.S84476. eCollection 2015. PMID 26396544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between the period of October, 2009 and August, 2011
Pre-assignment Details: Three patients were consented but not randomized due to failure to meet inclusion criteria (3 screen failures)
Groups:
- Lidocaine: Lidocaine will be infused through a catheter placed in the thoracic paravertebral space to block the transmission of pain signals at the level of the spinal nerves from the abdominal incision.
  At a concentration of 0.5%, Lidocaine has been deemed safe to use for peripheral nerve blocks and analgesia.Compared to ropivacaine, lidocaine is shorter-acting, less cardiotoxic, and safer to use.
  Lidocaine: Lidocaine will be infused through a catheter placed in the thoracic paravertebral space to block the transmission of pain signals at the level of the spinal nerves from the abdominal incision.
  At a concentration of 0.5%, Lidocaine has been deemed safe to use for peripheral nerve blocks and analgesia. There are several studies to support this as listed in the references. Compared to ropivacaine, lidocaine is shorter-acting, less cardiotoxic, and safer to use.
- Ropivacaine: Ropivacaine is a local anesthetic used as the standard drug in paravertebral nerve blocks at our institution. It is also used in other nerve block infusions at our hospital and institutions across the country. It will be used as the standard drug to which lidocaine is compared.
  Ropivacaine has been safely used in the paravertebral nerve blocks at our institution for several years.
  Ropivacaine: 0.5% Ropivacaine will be infused through a catheter placed in the thoracic paravertebral space to block the transmission of pain signals at the level of the spinal nerves from the abdominal incision. It is the local anesthetic used as the standard drug in paravertebral nerve blocks at our institution. It is also used in other nerve block infusions at our hospital and institutions across the country. It will be used as the standard drug to which lidocaine is compared.
Period: Overall Study
Arm/Group | Lidocaine | Ropivacaine
Started | 20 | 24
Completed | 17 | 18
Not Completed | 3 | 6
Not completed — Protocol Violation | 3 | 6

BASELINE CHARACTERISTICS:
Population: Patients undergoing elective laparoscopic bowel surgery with bilateral thoracic paravertebral continuous nerve blocks
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Ropivacaine | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Customized [Number; unit: participants]
  Age over 18 years | 17 | 18 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 8 | 16 | 24
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: 11-point Verbal Numerical Rating Scale (NRS) Pain Assessment
Description: The primary outcome of the study is the NRS score for pain at rest at 24 hours. The NRS Pain Assessment requires patients to select a number between 0 - 10 where 0 is no pain and 10 is the worst imaginable pain. Patients pick one whole number on this scale to describe their pain.
Time Frame: 24 hours from the end of surgery
Population: Patients undergoing elective laparoscopic bowel surgery with bilateral thoracic paravertebral continuous nerve blocks.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Lidocaine | Ropivacaine
Number analyzed (Participants) | 17 | 18
Scores on a scale | 3 [1 to 8] | 3 [3 to 8]

2. Secondary Outcome: Time to First Ambulation(Walking Greater Than 15 Feet)
Description: During the hospitalization following surgery until discharge. Hospital length of stay ranged from 3 - 22 days following surgery.
Time Frame: During the inpatient hospitalization (Hospital length of stay ranged from 3 - 22 days following surgery)
Population: 6 participants assigned to Group Ropi, 3 to Group Lido were not included in this analysis for the following reasons: 1 required mechanical ventilation post-op, 1 was excluded due to changes in surgical procedure, 2 patients did not complete PCA regimen, technical issues with block excluded 5 patients from analysis (considered protocol violations).
Measure: Median (Full Range); unit: days
Arm/Group | Lidocaine | Ropivacaine
Number analyzed (Participants) | 17 | 18
days | 2 [1 to 9] | 1 [1 to 22]
Statistical Analysis 1: Comparison: Lidocaine vs Ropivacaine; Test type: Non-Inferiority — A total sample size of 64 subjects (32 patients in each arm) is required to detect a difference of 0.5 SD, using an alpha error of 0.05 and a power of 0.8. After enrollment of 47 patients, we decided to complete the present interim analysis, and the study was then interrupted due to equivalence in results between the two groups; p = 0.148, t-test, 1 sided

3. Secondary Outcome: Time to First Flatus/Defecation
Description: as for outcome 2
Time Frame: During the inpatient hospitalization (Hospital length of stay ranged from 3 - 22 days following surgery)
Measure: Median (Full Range); unit: Postoperative days
Arm/Group | Lidocaine | Ropivacaine
Number analyzed (Participants) | 17 | 18
Postoperative days | 2 [1 to 3] | 2 [1 to 3]

4. Secondary Outcome: Hospital Length of Stay.
Description: as for outcome 2
Time Frame: During the inpatient hospitalization (Hospital length of stay ranged from 3 - 22 days following surgery)
Population: 6 participants assigned to Group Lopi, 3 to Group Lido were not included in this analysis for the following reasons: 1 required mechanical ventilation post-op, 1 was excluded due to changes in surgical procedure, 2 patients did not complete PCA regimen, and technical issues with block excluded 5 patients from analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Lidocaine | Ropivacaine
Number analyzed (Participants) | 17 | 18
days | 5 [4 to 9] | 5 [3 to 22]
Statistical Analysis 1: Comparison: Lidocaine vs Ropivacaine; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = .636, t-test, 1 sided

5. Secondary Outcome: Number of Patients With Complications (Including But Not Limited to Pneumonia, Atelectasis, Hypotension, Motor Weakness, Etc.)
Description: During the hospitalization following surgery until discharge.
Time Frame: During the inpatient hospitalization (Hospital length of stay ranged from 3 - 22 days following surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine | Ropivacaine
Number analyzed (Participants) | 17 | 18
Participants
  Hypotension (Patient 19) | 1 | 0
  Deydration with Acute Renal Failure (Patient 7) | 1 | 0
  Small Bowel Obstruction (Patients 43, 24, 34) | 1 | 2
  Rectal Bleeding (Patient 23) | 0 | 1
  Anastamotic Dehiscence with Pelvic Abscess -Pt. 34 | 0 | 1
  Tremors After Anesthetic Boli (Patient 34) | 0 | 1

6. Secondary Outcome: Postoperative Opioid Consumption (Milligrams of Dilaudid or Equivalent)
Description: as for outcome 2
Time Frame: During the inpatient hospitalization (Hospital length of stay ranged from 3 - 22 days following surgery)
Population: 6 participants assigned to Group Ropi, 3 to Group Lido were not included in this analysis for the following reasons: 1 required mechanical ventilation post-op, 1 was excluded due to changes in surgical procedure, 2 patients did not complete PCA regimen, and technical issues with block excluded 5 patients from analysis.
Measure: Mean (Full Range); unit: Milligrams
Arm/Group | Lidocaine | Ropivacaine
Number analyzed (Participants) | 17 | 18
Milligrams
  Hydromorphone PACU | 1.6 [0 to 14.4] | 1.1 [0.2 to 8.3]
  Hydromorphone 24HRS | 9.2 [1.2 to 29.3] | 5.7 [1.4 to 24.2]
  Hydromorphone 48HRS | 16.1 [1.6 to 54.7] | 9.6 [2 to 39.5]
Statistical Analysis 1: Comparison: Lidocaine vs Ropivacaine; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.193, t-test, 2 sided — Hydromorphone consumption (mg) in Post-Anesthesia Care Unit (PACU)
Statistical Analysis 2: Comparison: Lidocaine vs Ropivacaine; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.635, ANOVA — Hydromorphone consumption (mg) in PACU versus at 24 hours versus 48 hours

7. Secondary Outcome: Consumption of Nerve Block Boluses Will Also be Recorded Daily
Description: During the hospitalization following surgery until discontinuation of the block or discharge. Hospital length of stay ranged from 3 - 22 days following surgery.
Time Frame: During the inpatient hospitalization (Hospital length of stay ranged from 3 - 22 days following surgery)
Population: as for outcome 4
Measure: Median (Full Range); unit: milliliters
Arm/Group | Lidocaine | Ropivacaine
Number analyzed (Participants) | 17 | 18
milliliters
  Nerve block boluses PACU | 20 [0 to 40] | 20 [0 to 40]
  Nerve block boluses 24HRS | 0 [0 to 12] | 0 [0 to 30]
  Nerve block boluses 48HRS | 0 [0 to 6] | 0 [0 to 18]
Statistical Analysis 1: Comparison: Lidocaine vs Ropivacaine; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.063, ANOVA; Local Anesthetic Consumption through para-vertebral catheters in PACU vs. at 24 hours vs. 48 hours

ADVERSE EVENTS:
Arm/Group | Lidocaine | Ropivacaine
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 1/17 | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=17) | Ropivacaine (N=18)
Surgical Complications (Surgical and medical procedures) | 1 (1) | 4 (4) — Five patients reported surgical complications including dehydration with acute renal failure, small bowel obstruction, rectal bleeding, and anastomotic dehiscence with pelvic abscess. Further separation of is not possible.

LIMITATIONS AND CAVEATS:
This study did not provide information about the treatment drug mechanism of action, whether it is regional or systemic. Local anesthetic plasma concentration was not measured in this study either.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No